CLINICAL TRIAL: NCT02525965
Title: The Influence of Resection Margin on the Recurrence of Early-stage Hepatocellular Carcinoma After Hepatectomy: a Randomized Controlled Trial
Brief Title: The Influence of Resection Margin on the Recurrence of Early-stage Hepatocellular Carcinoma
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Eastern Hepatobiliary Surgery Hospital (Other)
Responsible Party: Principal Investigator, ShenFeng, vice president of the Eastern Hepatobiliary Surgery Hospital, Eastern Hepatobiliary Surgery Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: EHBHLRM-2015-8-10
Record Dates: First submitted 2015-08-10; First posted 2015-08-18 (Estimated); Last update posted 2016-03-31 (Estimated); Status verified 2016-03

CONDITIONS: Hepatocellular Carcinoma
Keywords: Wide resection margin; Recurrence; Early-stage hepatocellular carcinoma
MeSH Terms: conditions — Carcinoma, Hepatocellular; Recurrence

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Wide resection margin >1cm (Experimental): Surgical removal of lesions choosing the method of wide resection margin >1cm
  Interventions: Procedure: Wide resection margin >1cm
- Narrow resection margin <1cm (Active Comparator): Surgical removal of lesions choosing the method of narrow resection margin <1cm
  Interventions: Procedure: Narrow resection margin <1cm

INTERVENTIONS:
Procedure: Wide resection margin >1cm — Surgical removal of lesions choosing the method of wide resection margin >1cm
  Arms: Wide resection margin >1cm
Procedure: Narrow resection margin <1cm — Surgical removal of lesions choosing the method of wide resection margin <1cm
  Arms: Narrow resection margin <1cm

SUMMARY:
Before the surgery, the investigators predict the risk of microvascular invasion (MVI) presence for the early-stage hepatocellular carcinoma according to the nomogram the investigators have created. Patients with a high risk of microvascular invasion were randomly chose to give the treatment of a wide resection margin, which establish an individualized anti-recurrence program based on the high-grade evidence-based medicine.

DETAILED DESCRIPTION:
Although liver resection is still the first line of treatment for hepatocellular carcinoma (HCC) presently, 5-year overall recurrence rates > 70%, the same with early-stage hepatocellular carcinoma, for some studies reported the rates > 40%. Recurrence is also the first cause of death in these patients, so recurrence is the most important factors affecting surgical results of HCC. For the precaution of cancer recurrence, there are no proven techniques for clinical reference at present.

For now, there has been many controversies on the impact about the width of liver resection margin on curative effect. Poon has proven that there is no significant difference in recurrence rate between resection margin > 1cm and resection margin < 1cm. However, Shi et al published a randomized controlled trial: for patients with a solitary tumor, resection margin > 2cm can reduce the recurrence rate after hepatectomy. This is also the only randomized clinical trial study which proves increaseing resection margin will benefit the clinical results at present. A meta analysis consist of 18 studies proves that whether the resection margin has a relationship with a benefit clinical result still needs a further verification.

On the other hand, because microvascular invasion (MVI) is the direct evidence of the micro metastasis in hepatocellular carcinoma, it will decrease recurrence rate for the patients with a high MVI risk, if the investigators increase the resection margin width during the surgery? Shanghai Eastern Hepatobiliary Surgery Hospital which the investigators affiliated with had ever conducted a retrospective analysis on consecutive 3263 patients with HCC hepatectomy, the results indicated that a wide resection margin（≥1cm）can benefit those patients with microvascular invasion , nevertheless, the benefit will not present if patients are without microvascular invasion.

Further and better proofs still needs to approval this consequence, of course. In the past，another study of the ours, published online in the Journal of the American Medical Association Surgery, established a nomogram to predict the presence of microvascular invasion in the early-stage hepatocellular carcinoma, it will efficiently predict the occurrence of microvascular invasion in the hepatocellular carcinoma (HCC) fulfilled the Milan criteria. In consideration of the above basis, the investigators will implement a randomized controlled trial to certificate whether it could really reduce the recurrence rate after liver resection for participants with a high MVI risk during the surgery, if the method participants chose is a wide resection margin.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients > 18 years and <=70 years of age.
* Diagnosed with HCC according to the criteria of American Association for the Study of Liver Diseases (AASLD).
* Fulfill the Milan criteria.
* High-risk of microvascular invasion (MVI).
* Nomogram score >200.
* Performance status score is 0-1 before the surgery.
* Without or mild liver cirrhosis and the liver function is Child A class.
* Without any other treatments such as TACE、PEI、PRFA before the surgery.

Exclusion Criteria:

* Patients with macro tumor thrombus or extrahepatic metastasis.
* Patients with apparent cardiac, pulmonary, cerebral and renal dysfunction.
* Subjects accepting other trial drugs or participating in other clinical trials.
* Patients refuse to join our trial.
* Female with pregnancy or during the lactation period.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 194 (Estimated)
Dates: Start 2015-08; Primary Completion 2017-12 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Overall survival rates of each group | 3 years

SECONDARY OUTCOMES:
Occurrence rate of recurrence of each group | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Shen Feng, MD, Study Chair — Eastern Hepatobiliary Surgery Hospital, Second Military Medical University
Locations (1):
- Eastern hepatobilliary surgery hospital, Shanghai, Shanghai Municipality, China